CLINICAL TRIAL: NCT07394166
Title: Brief Tech-Parenting for Regulatory Screen Use in Young Children: A Pilot Study
Brief Title: Balancing Emotions and Electronics: A Pilot Intervention for Preschoolers
Acronym: BEE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Virginia Peisch, Instructor of Pediatrics, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00052998
Record Dates: First submitted 2026-01-05; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Screen Media Use
Keywords: childhood; screen time; parenting; intervention; self-regulation; preschool
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): 3-session, virtual group therapy
  Interventions: Behavioral: Brief-RSU

INTERVENTIONS:
Behavioral: Brief-RSU — Brief-RSU Intervention: The Brief-RSU intervention consists of three, 60-minute sessions, outlined in Table 1. Brief-RSU aims to reduce RSU while increasing adaptive caregiver tools. Treatment targets include: 1) psychoeducation, 2) scheduling screen time to consistent times, 3) "planning ahead" for times when RSU is likely to occur, and 4) teaching the RULER approach[9, 10] to strengthen caregiver socialization of child emotion regulation (replacement behavior).

SUMMARY:
This study is testing a brief, virtual therapy for caregivers of preschool children. The goal is to reduce use of screen time to regulate young children's emotions and boredom, i.e. "regulatory screen use" (RSU). We expect that RSU negatively impacts young children's ability to cope with emotions and boredom. Thus, reducing RSU should improve children's self-regulation. The intervention will include three, 60-minute group sessions with caregivers, and remote data collection at three time points (pre-intervention, post-intervention, and 1-month follow-up).

DETAILED DESCRIPTION:
Project Aims / Hypotheses. This intervention study aims to refine and test a brief, caregiver delivered therapeutic program targeting the problematic use of screen time to regulate young children's emotions and boredom, i.e. "regulatory screen use" (RSU). RSU is a candidate mechanism for the negative impacts of screen time on children's mental health; therefore, this proposal addresses the growing public health concern related to pervasive digital media use. Our group has already developed an effective brief tech-parenting program for school-age children; the current study will expand this intervention to target RSU in young children.

Aim 1: Develop and test the acceptability and feasibility of a brief tech-parenting intervention targeting RSU (Brief-RSU) with caregivers of 30 children ages 30-54 months. Hypothesis 1: We expect that Brief-RSU will be highly acceptable and feasible, as evidenced by high retention rates and positive caregiver feedback.

Aim 2: Determine the efficacy of Brief-RSU on caregiver and child outcomes. We expect that Brief-RSU will increase adaptive caregiving (e.g., emotion coaching; reduction in RSU) from pre to post (Hypothesis 2a) and significantly improve child emotion and behavior regulation (Hypothesis 2b).

Background. Significant concern among scientists and the public has emerged over the last decade regarding the adverse effects of screen media activity on child development, including poor sleep, reduced educational achievement, greater behavior problems, inattention, and anxiety. Despite this widespread concern, clinical recommendations on child digital media management are currently lacking, primarily due to gaps in our knowledge base. Existing research predominantly relies on simplistic screen media measures, such as total screen time, that do not consider the context and function of screen media use. Altogether, there is an urgent need to expand what is known about the mechanisms by which digital media negatively impact child development in order to provide effective and evidence-based recommendations to caregivers, clinicians, and policymakers.

Regulatory screen use (RSU), which describes the use of screen media to calm or occupy children at home and in public, has already been shown to be highly prevalent and associate with poor child outcomes. For example, a longitudinal study of more than 400 preschoolers found that higher RSU at baseline predicted worse executive functioning in girls and more emotional reactivity in boys 6 months later. Further, a study of 200 preschool-age children found concurrent associations between RSU, empathy, and emotional control. We propose that RSU affects psychosocial development by depriving children of critical opportunities to practice self-regulation skills. The proposed study will be the first to test whether a brief, caregiver-focused intervention can reduce RSU, while also strengthening adaptive parenting and child emotional well-being.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver endorses regulatory screen use
* Child age 30-54 months at enrollment
* English speaking

Exclusion Criteria:

* Intellectual disability or global developmental delay
* Autism spectrum disorder
* Child in the custody of DCF

Ages: 30 Months to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-26 (Estimated)

PRIMARY OUTCOMES:
Regulatory Screen Use (RSU) | Baseline; 1-month follow up (i.e., 1 month after the last workshop).
  Caregiver reported frequency of using screen time and non-screen time strategies to regulate a child's emotions. For example, the caregiver is asked how frequently they use screens (e.g., iPad; smartphone) to help keep their child calm when they are expected to sit still (e.g., at a restaurant). Seven different situations/settings are assessed (e.g., sibling conflict; at church or doctor's office).

SECONDARY OUTCOMES:
Child self-regulation (BRIEF-Preschool) | Baseline; 1-month follow up (i.e., 1 month after the last workshop).
  Caregiver report on an age- and gender-normed questionnaire assessing child emotional and behavioral regulation.
Parental Stress Scale | Baseline; 1-month follow up (i.e., 1 month after the last workshop).
  Caregiver self-report of confidence and stress related to parenting. The caregiver is asked to select one option (1=strongly disagree; 5=strongly agree) on questions related to their experience parenting. There is a total of 18 questions.
Perceived Stress Scale | Baseline; 1-month follow up (i.e., 1 month after the last workshop).
  Caregiver self-report of general stress and well-being. The caregiver is asked to select one response option (0=never; 4=very often) that best describes their current level of perceived stress. There is a total of 10 questions.

OTHER OUTCOMES:
Acceptability of Workshop | Immediately following the 3-session workshop.
  After completion of the three workshops on RSU, participant will be asked to provide feedback on how helpful the workshop curriculum was and how much they learned (managing child screen time; regulating their child's emotions).

IPD SHARING:
Plan to Share IPD: Undecided
Limited IPD will be shared upon reasonable request from the researcher.